CLINICAL TRIAL: NCT04228224
Title: Stroke Rehabilitation Program Based on a Powered Lower Extremity Exoskeleton in Chile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporación de Rehabilitación Club de Leones Cruz del Sur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CorporacionRCLCS0001
Record Dates: First submitted 2020-01-08; First posted 2020-01-14 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Stroke; Hemiparesis; Gait; Brain-Computer Interface; Rehabilitation; Exoskeleton
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robot-assisted Rehabilitation (Experimental): Participants will receive Robot-assisted training with a lower extremity powered exoskeleton (H3 Exoskeleton, Spain). Patients will perform lower limb exercises assisted by the device. Training involve 24 sessions, 2 sessions per week for 12 weeks, each lasting about 1 hour.
  Interventions: Device: Robot-assisted training with a lower extremity powered exoskeleton (H3 Exoskeleton, Spain)
- Conventional Gait Rehabilitation (Active Comparator): Participants in this group will perform conventional gait rehabilitation on a rehabilitation institution with assistance of a physical therapist. Training involve 24 sessions, 2 sessions per week, each session lasting about 1 hour.
  Interventions: Behavioral: Conventional gait rehabilitation

INTERVENTIONS:
Device: Robot-assisted training with a lower extremity powered exoskeleton (H3 Exoskeleton, Spain) — The H3 is a powered lower extremity exoskeleton with actuated at hips, knees and ankles joints. A novel control software has been design and implemented in this device, which allows selective joint movement and recording of data from each rehabilitation session.
  Arms: Robot-assisted Rehabilitation
Behavioral: Conventional gait rehabilitation — Conventional gait rehabilitation consist in walking and other applicable lower limb exercises performed by participants with assistance of a physical therapist.
  Arms: Conventional Gait Rehabilitation

SUMMARY:
This research will study the effects of a rehabilitation program assisted by a powered lower extremity exoskeleton in patients after stroke. It will compare clinical and biomechanical features of patients at baseline and after intervention. Additionally, it will also examine the use of a brain-computer-interface (BCI) to command movements on the powered lower limb exoskeleton. The findings will be used to improve understanding human-robot interaction, to improve the design of the robotic devices and to improve rehabilitation services.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of mortality, morbidity and disability in adults in developed countries. Survivors may suffer several neurological deficits or deficiencies, such as hemiparesis, communication disorders, cognitive deficits and visuospatial perception disorders. Hemiplegia is a par loss of hemi-body voluntary motricity following a brain injury, usually resulting in alterations of the locomotor system with persistent disorders of movement and posture. Hemiplegia significantly affects gait performance. Gait recovery is an important objective in the rehabilitation program for stroke patients.The currently available treatment techniques include classical techniques of gait rehabilitation, functional electrical stimulation, electromechanic devices, robotic devices and brain-computer interfaces, among others.The evidence suggest that the combination of different rehabilitation strategies is more effective than conventional rehabilitation techniques alone. Technology-based rehabilitation methods such as robotic devices need more research to demonstrate their effects on gait recovery.

This study will assess the effects of a rehabilitation program with a powered lower extremity exoskeleton in people with stroke. Additionally, it will also examine the use of a brain-computer-interface (BCI) to command movements on the powered lower limb exoskeleton. The findings will be used to improve understanding human-robot interaction, to improve the design of the robotic devices and to improve rehabilitation services.

ELIGIBILITY:
Inclusion Criteria:

* unilateral lower extremity paresis
* haemorrhagic or ischemic stroke
* a minimum of six months after the acute infarction/onset of the disease
* full passive range of motion in lower extremity or at least at neutral position
* be able to stand freely
* be able to walk with or without aid for at least 20 meters in less than 2 minutes

Exclusion Criteria:

* peripheral nervous system pathology
* epilepsy
* weight over 100 kg
* no cognitive ability to follow the study instructions
* pregnancy
* use of implanted devices
* instable lower extremity joints or fixed contracture

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Gait Deviation Index Baseline | Baseline
  Gait Deviation Index will be calculated for each patient using a 3D VICON infra-red camera system.
Gait Deviation Index Post-Intervention | 12 weeks
  Gait Deviation Index will be calculated for each patient using a 3D VICON infra-red camera system.

SECONDARY OUTCOMES:
Maximal muscle strength Baseline | Baseline
  Maximal muscle strength (peak torque, Nm) during maximal voluntary unilateral hip extension-flexion, and hip adduction-abduction (standing), knee extension-flexion (seated), respectively. Both the affected (AF) and non-affected (NA) leg. A hand-held dynamometer will be used for the assessment.
Maximal muscle strength Post-Intervention | 12 weeks
  Maximal muscle strength (peak torque, Nm) during maximal voluntary unilateral hip extension-flexion, and hip adduction-abduction (standing), knee extension-flexion (seated), respectively. Both the affected (AF) and non-affected (NA) leg. A hand-held dynamometer will be used for the assessment.
Distance in 6 Minute Walk Test (6MWT) Baseline | Baseline
  Measure of the distance a subject covers during an indoor gait on a flat, hard surface in 6 minutes, using assistive devices, as necessary. The test consist in a evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance.
Distance in 6 Minute Walk Test (6MWT) Post-Intervention | 12 weeks
  Measure of the distance a subject covers during an indoor gait on a flat, hard surface in 6 minutes, using assistive devices, as necessary. The test consist in a evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance.
Muscle tone measured using modified ashworth scale (MAS) Baseline | Baseline
  Tests resistance to passive movement about a joint with varying degrees of velocity. A score of 1 indicates no resistance, and 5 indicates rigidity.
Muscle tone measured using modified ashworth scale (MAS) Post-Intervention | 12 weeks
  Tests resistance to passive movement about a joint with varying degrees of velocity. A score of 1 indicates no resistance, and 5 indicates rigidity.
Passive range of motion Baseline | Baseline
  Passive range of motion in lower extremities. ROM will be assessed by using an universal goniometer
Passive range of motion Post-Intervention | 12 weeks
  Passive range of motion in lower extremities. ROM will be assessed by using an universal goniometer
10 meter walk test Baseline | Baseline
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
10 meter walk test Post-Intervention | 12 weeks
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
Timed Up and Go Baseline | Baseline
  Measurement of the time in seconds for a person to rise from sitting from a standard arm chair, walk 3 meters, turn, walk back to the chair, and sit down. The person wears regular footwear and customary walking aid.
Timed Up and Go Post-Intervention | 12 weeks
  Measurement of the time in seconds for a person to rise from sitting from a standard arm chair, walk 3 meters, turn, walk back to the chair, and sit down. The person wears regular footwear and customary walking aid.
Berg Balance Scale Baseline | Baseline
  Berg balance scale is used for functional balance. participants are asked to perform 14 tasks frequently used in daily life activities. The highest possible score is 56 points. A higher score indicates better balance.
Berg Balance Scale Post-Intervention | 12 weeks
  Berg balance scale is used for functional balance. participants are asked to perform 14 tasks frequently used in daily life activities. The highest possible score is 56 points. A higher score indicates better balance.
Functional Ambulation Classification (FAC) Baseline | Baseline
  FAC is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
Functional Ambulation Classification (FAC) Post-Intervention | 12 weeks
  FAC is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
Patient satisfaction with device: Quebec User Evaluation of Satisfaction with Assistive Technology | 12 weeks
  Measured with QUEST scale. The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) is a 12-item outcome measure that assesses user satisfaction with two components, Device and Services. Scores of 1 indicate dissatisfaction and scores of 5 indicate high satisfaction
Medical Research Council test (MRC) Baseline | Baseline
  Manual evaluation of muscle strength. This scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle. Grade 0 = no movement is observed, grade 5= muscle contracts normally against full resistance. Six muscles groups are tested at both sides of the body: shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, ankle dorsiflexion. Maximal total score is 60.
Medical Research Council test (MRC) Post-Intervention | 12 weeks
  Manual evaluation of muscle strength. This scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle. Grade 0 = no movement is observed, grade 5= muscle contracts normally against full resistance. Six muscles groups are tested at both sides of the body: shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, ankle dorsiflexion. Maximal total score is 60.
Gait Speed Baseline | Baseline
  Gait Speed will be calculated for each patient using a 3D VICON infra-red camera system.
Gait Speed Post-intervention | 12 weeks
  Gait Speed will be calculated for each patient using a 3D VICON infra-red camera system.

CONTACTS AND LOCATIONS:
Overall Officials: Asterio H Andrade Gallardo, MSc., Study Chair — Corporación de Rehabilitacion Club de Leones Cruz del Sur
Locations (1):
- Corporación de Rehabilitación Club de Leones Cruz del Sur, Punta Arenas, Region of Magallanes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flansbjer UB, Holmback AM, Downham D, Patten C, Lexell J. Reliability of gait performance tests in men and women with hemiparesis after stroke. J Rehabil Med. 2005 Mar;37(2):75-82. doi: 10.1080/16501970410017215. PMID 15788341
- [Background] Belda-Lois JM, Mena-del Horno S, Bermejo-Bosch I, Moreno JC, Pons JL, Farina D, Iosa M, Molinari M, Tamburella F, Ramos A, Caria A, Solis-Escalante T, Brunner C, Rea M. Rehabilitation of gait after stroke: a review towards a top-down approach. J Neuroeng Rehabil. 2011 Dec 13;8:66. doi: 10.1186/1743-0003-8-66. PMID 22165907
- [Background] Bortole M, Venkatakrishnan A, Zhu F, Moreno JC, Francisco GE, Pons JL, Contreras-Vidal JL. The H2 robotic exoskeleton for gait rehabilitation after stroke: early findings from a clinical study. J Neuroeng Rehabil. 2015 Jun 17;12:54. doi: 10.1186/s12984-015-0048-y. PMID 26076696
- [Background] Wallard L, Dietrich G, Kerlirzin Y, Bredin J. Effects of robotic gait rehabilitation on biomechanical parameters in the chronic hemiplegic patients. Neurophysiol Clin. 2015 Sep;45(3):215-9. doi: 10.1016/j.neucli.2015.03.002. Epub 2015 Sep 14. PMID 26381192